CLINICAL TRIAL: NCT00235482
Title: Intratumoural Administration of Coxsackievirus A21 for the Control of Malignant Melanoma (PXS-X02)
Acronym: PXS-X02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viralytics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V937-002; PSX-X02 (Other: Viralytics Study ID)
Record Dates: First submitted 2005-10-07; First posted 2005-10-10 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: CAVATAK

INTERVENTIONS:
Drug: Coxsackievirus A21

SUMMARY:
The purpose of this study is to determine the safety of an injection of coxsackievirus A21 into a melanoma tumour, and also to see if there is a tumour response.

DETAILED DESCRIPTION:
Coxsackievirus A21, a naturally occurring enterovirus, has shown that in vivo it can infect and lyse melanoma. This study is to assess safety of a single intratumoural injection of the virus into an accessible subcutaneous melanoma metastasis.

ELIGIBILITY:
Inclusion Criteria:

* stage IV melanoma (AJCC classification)
* minimum of 2 sc metastases
* failure or refusal of standard chemotherapy
* ECOG score of 0 or 1
* other

Exclusion Criteria:

* metastatic CNS disease
* ocular or mucosal melanoma
* immunodeficiency
* splenectomy
* other

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-11-08 (Actual); Primary Completion 2006-04-21 (Actual); Study Completion 2006-04-21 (Actual)

PRIMARY OUTCOMES:
Safety profile of treatment, characterisation of adverse events

SECONDARY OUTCOMES:
Efficacy - clinical response of injected and non-injected tumours

CONTACTS AND LOCATIONS:
Locations (1):
- Melanoma Unit, Mater Misericordiae Hospital, Newcastle, New South Wales, Australia